CLINICAL TRIAL: NCT00972907
Title: An Open Label Study to Examine the Effect of Coated Nifedipine Suppository on Anal Fissure Pain and Healing in Human Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Nir Barak MD, RDD Pharma LTD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDD 104
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Anal Fissure
Keywords: anal fissure; pain; nifedipine
MeSH Terms: conditions — Fissure in Ano; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Nifedipine coated suppositories BID.
  Interventions: Drug: Nifedipine coated suppositories

INTERVENTIONS:
Drug: Nifedipine coated suppositories — 12 mg Nifedipine coated suppositories BID

SUMMARY:
This is an open label study. The study will consist of 1 treatment group: coated Nifedipine suppository containing 12 mg of Nifedipine, administered BID to subjects with chronic anal fissure.

DETAILED DESCRIPTION:
This is an open label study. The study will consist of 1 treatment group: coated Nifedipine suppository containing 12 mg of Nifedipine. Approximately 20 subjects will participate into this 8-week study. A screening visit will be used to determine subject suitability for inclusion in the trial. Within one week of the screening visit, subjects who meet all inclusion criteria and none of the exclusion criteria will receive Coated Nifedipine 12 mg Suppository X2 a day (BID) (24 mg/day total) for a period of 8 weeks. During this period, 4 study visits (at 0, 2, 5, and 8 weeks) will take place. Study medication will be administered BID (in the morning and in the evening). In addition to receiving study medication, subjects will be maintained on a standard treatment for Anal Fissure: sitz baths, high fiber diet.

ELIGIBILITY:
Inclusion Criteria:

* Single anal fissure
* Signed written informed consent
* Male or female subjects 18 to 65 years of age
* Has chronic anal fissure defined as history of anal pain at least three days a week for 30 days duration or more
* Visible fibers of the internal sphincter were seen at the base of the fissure or if a sentinel pile was present
* VAS of > 35 mm in screening visit
* If female, is nonlactating, has a negative urine pregnancy test result, and does not plan on becoming pregnant during the study, or not of childbearing potential (hysterectomy or tubal ligation at least 6 months prior to entry to the study or post-menopausal for 1 year); if of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice or be willing to continue to practice appropriate birth control (such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire study duration.

Exclusion Criteria:

* Known allergy to Nifedipine, polyethylene-glycol, propylene Glycol or silicone
* Fissure resulting from inflammatory bowel disease, venereal disease, perianal psoriasis, immunodeficiency syndrome
* Anal abscess
* Fixed anal stenosis
* Active or past history of cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, moderate to severe congestive heart failure, or cardiac valve abnormalities
* Type 1 diabetes mellitus
* Insulin treated type 2 diabetes mellitus
* History of Renal insufficiency
* History of Liver insufficiency
* Malignant disease within 5 years of screening
* Has uncontrolled hypertension (sitting blood pressure <160/95 mmHg at screening)
* History of chronic gastrointestinal disease
* History of rectal surgery
* History of gastrointestinal surgery
* History of HIV, hepatitis B, hepatitis C
* In need of chronic use of medication, with the exception of birth control medications
* Currently uses medication for acute illness (other than medications for use of treatment/pain relief of anal fissure)
* Has used, in the last four weeks, drugs that may affect blood coagulation, such as Aspirin at a dose higher than 500 mg/day , Warfarin, Sintrom, Enoxaparin, Nadroparin, Heparin, Clopidogrel, Ticlopidine
* Is using drug that may affect rectal tone
* Calcium Channel Blocker such as:

  * Nifedipine (Osmo-Adlat, Pressolat, Nifedipine -Teva, Nifedilong)
  * Amlodipine (Amlow, Norvasc, Amlodipine-Teva)
  * Lercadipine (Vasodip)
  * Verapamil (Ikacor, Ikapress, Verapress)
  * Felodipine (Penedil)
  * Diltiazem (Adizem, Dilatam)
* Nitrate donors such as:

  * Glyceryl Trinitrate (Deponit)
  * Isosorbid dinitrate (Isoket, Isolong)
  * Isosrbid mononitrate (Monocord, Monolong, Mononit)
  * Nitroglycerine (Nitrocine, Nitroderm, Nitrolingual)
* Has upon physical examination a rectal deformation or signs of rectal disease such as bleeding hemorrhoids, fistula., infection or space occupying lesion
* Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site; or is employed by RDD Pharma Ltd

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To examine the effect of coated Nifedipine suppository on Anal fissure pain. | 8 weeks
To examine the effect of coated Nifedipine suppository on Anal fissure healing. | 8 weeks

SECONDARY OUTCOMES:
To investigate the Safety and tolerability of coated Nifedipine suppositories in Anal Fissure patients. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sapir Medical Center, Kfar Saba
  - Macabi HMO, Tel Aviv